CLINICAL TRIAL: NCT07183722
Title: Clinical and Biological Impact of Gut Microbiota on the Development of Bacteremia and Outcomes in Adult Patients With Bacteremia During the COVID-19 Pandemic
Brief Title: Clinical and Biological Impact of Gut Microbiota in Adult Patients With Bacteremia During the COVID-19 Pandemic
Acronym: SURVEIL
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.Microb.22.01
Record Dates: First submitted 2025-09-03; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — rectal swab, nasopharyngeal swab, and peripheral blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Microbiota analysis — Analysis of microbiota in patients admitted to the following departments: General Anesthesia and Resuscitation, Cardio-Thoracic-Vascular Anesthesia and Resuscitation, Internal Medicine, and MeCAU.

SUMMARY:
The widespread use of antibiotics in healthcare, veterinary, and agricultural sectors has significantly contributed to the rise of antimicrobial resistance (AMR), affecting both commensal and pathogenic microorganisms. AMR infections are linked to poorer patient outcomes, prolonged hospital stays, and increased mortality. The COVID-19 pandemic exacerbated this issue through the overuse of antibiotics in hospitalized patients, worsening global resistance trends. Six bacterial species-Enterococcus faecium, Staphylococcus aureus, Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa, and Enterobacter spp.-are considered urgent targets for new drug development. Advanced diagnostic methods, particularly Next Generation Sequencing (NGS), show promise in improving the detection and management of sepsis and resistant infections. However, effective application of NGS requires interdisciplinary collaboration and specialized expertise, highlighting the need for integrated efforts between research institutions and clinical centers to improve AMR surveillance, diagnostics, and treatment strategies.

DETAILED DESCRIPTION:
Excessive consumption of antibiotics in clinical, veterinary, and agricultural settings has led to a huge influx of antibiotics into the environment. This has driven the evolution of antimicrobial resistance (AMR) in commensal and pathogenic microorganisms.

Infections related to AMR microorganisms are associated with an increased incidence of negative outcomes for patients, longer hospital stays, and higher morbidity and mortality rates.

A list of six bacterial species has been drawn up for which it is mandatory to discover and develop new drugs: Enterococcus faecium, Staphylococcus aureus, Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa, and Enterobacter spp.

The pandemic has led to an exponential increase in the use of antibiotics in hospitalized COVID-19 patients, resulting in increased antibiotic resistance and a worsening of the global epidemiological picture.

Laboratories are focusing on certain multi-resistant microorganisms (MDR) such as A. baumannii, P. aeruginosa, K. pneumoniae, and E. coli, considered critical priorities by the World Health Organization (WHO), but Staphylococcus aureus and Enterococcus fecium also continue to pose a problem in the management of patients admitted to intensive care. Faced with this critical issue, there is an increasingly urgent need for new and more effective diagnostic and therapeutic tools capable of controlling its spread. Data collection, as well as analysis of the impact that the pandemic has had on AMR, is essential for implementing surveillance, monitoring, and control systems.

The most studied diagnostic pathway in infectious diseases is that of the septic patient, as sepsis is the most serious complication of any infection, even minor ones. Sepsis is difficult to diagnose and must be treated promptly.

The implementation of Next Generation Sequencing (NGS) technologies in infectious diseases is also very promising in the field of sepsis diagnostics, as well as in the study of SARS COV-2 variants, microbiota, and bacterial resistance. However, it requires clinical microbiological and bioinformatic know-how to interpret and evaluate NGS data and place this data in the appropriate clinical context. For this reason, scientific collaboration between universities and hospitals is crucial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients admitted to the following departments: General Anesthesia and Resuscitation, Cardio-Thoracic-Vascular Anesthesia and Resuscitation, Internal Medicine, and MeCAU
* Signature of informed consent to participate in the study.

Exclusion Criteria:

• Absence of informed consent signature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the following departments: General Anesthesia and Resuscitation, Cardio-Thoracic-Vascular Anesthesia and Resuscitation, Internal Medicine, and MeCAU.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Microbiota Analysis | Through study completion, an average of 1 year
  Studying the gut microbiota of patients colonized/infected with multidrug-resistant microorganisms to assess the potential role of protective factors against colonization and bacteremia caused by these microorganisms.

SECONDARY OUTCOMES:
Analysis of genetic variants | Through study completion, an average of 1 year
  Minimum number of genetic variants characterizing resistance to new drugs, also for the purpose of developing rapid investigation systems for early monitoring.
Phylogenetic correlation of genomic resistance profiles | Through study completion, an average of 1 year
  Phylogenetic correlation of genomic resistance profiles, using NGS techniques and bioinformatic processing, of strains isolated during hospitalization;
Antibiotic susceptibility | Through study completion, an average of 1 year
  Antibiotic susceptibility of E. coli, K. pneumoniae, P. aeruginosa, and A. baumannii to the new drugs cefiderocol and fosfomycin
Identify the optimal model for rapid diagnosis | Through study completion, an average of 1 year
  Identify the optimal model for rapid diagnosis, including from an economic standpoint, comparing the organizational models and fast track pathways for bacteremia of two italian University Hospital

CONTACTS AND LOCATIONS:
Locations (1):
- SSD Laboratori di Ricerca (DAIRI) - AOU Alessandria, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: No